CLINICAL TRIAL: NCT03934723
Title: Do Antidepressant Medications Blunt Responses to Exercise Training in Overweight and Obese Individuals?
Brief Title: Does Antidepressant Use Blunt Adaptations to Exercise?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: California State University, San Marcos (Other)
Responsible Party: Principal Investigator, Matthew Schubert, Assistant Professor of Kinesiology, California State University, San Marcos
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1423972-1
Record Dates: First submitted 2019-04-26; First posted 2019-05-02 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Depression; Depressive Disorder; Metabolic Syndrome
Keywords: Exercise; Antidepressants; Visceral fat
MeSH Terms: conditions — Depression; Depressive Disorder; Metabolic Syndrome; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): This arm will consist of healthy overweight and obese individuals who are physically inactive and do not have clinically diagnosed depression or depression symptoms.
  Interventions: Behavioral: Exercise
- Antidpressants (Experimental): This arm will consist of healthy overweight and obese adults who are physically inactive and who are diagnosed with clinical depression and have been taking antidepressant medications for at least 1 year.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — The intervention consists of 180 minutes of moderate-vigorous aerobic exercise per week for 6 weeks.

SUMMARY:
Nearly one out of ten US adults over the age of 18 currently takes antidepressant medication, which can also treat other conditions such as anxiety. Combining pharmaceutical treatment with exercise may yield even greater benefits than using drugs alone, and this is commonly prescribed for depression. However, little is known about the drug-exercise interactions and their influence on metabolic health. A common side effect of antidepressant use is weight gain, particularly abdominal (visceral) fat, which is highly detrimental to overall health. Exercise is a well-known counter to abdominal fat accumulation. The aim of the proposed study is to compare the efficacy of 6 weeks of exercise training to reduce abdominal fat in healthy overweight/obese adults either taking or not taking antidepressant medication. Twenty-four inactive overweight/obese, but otherwise healthy, adults will complete 6 weeks of an exercise training intervention consisting of three days of aerobic exercise training per week. Participants will either not be taking antidepressant medication or will have been on their medication for at least 1 year. The primary outcome will be abdominal fat determined by waist circumference and dual x-ray absorptiometry, which is considered one of the optimal methods for assessment of abdominal fat.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be English language speakers
* Male or females between the ages of 18-40.
* All genders and ethnicities.
* Healthy as assessed by a health history questionnaire (no diagnosed physical diseases or conditions preventing participation in exercise).
* Individuals on antidepressants will be recruited if they are consuming selective serotonin reuptake inhibitors (SSRIs) and selective serotonin and norepinephrine reuptake inhibitors (SNRIs) only. Participants will send prescription information after consent has been provided as part of the screening process, including the dose and frequency of medication.
* A body mass index (BMI) of 25 or greater is required for inclusion.

Exclusion Criteria:

* Inability to complete moderate-vigorous exercise.
* Taking first generation antidepressant medications or other medications such as monoamine oxidase inhibitors (MAOI).
* Other medications, such as medications for attention-deficit hyper-activity disorder or metabolism
* Undiagnosed depression that may be unveiled during the screening process.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-06-15 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Visceral adipose tissue (VAT) | Change from baseline after 6 weeks.
  VAT assessed by dual-energy X-ray absorptiometry (DXA)
Waist circumference | Change from baseline after 6 weeks.
  Waist circumference is a proxy of VAT

SECONDARY OUTCOMES:
Aerobic fitness | Change from baseline after 6 weeks.
  Fitness assessed via a maximal treadmill exercise test
Blood pressure | Change from baseline after 6 weeks.
  Resting blood pressure assessed with an oscillatory blood pressure monitor
Blood glucose | Change from baseline after 6 weeks.
  Fasting capillary glucose sample
Blood lipid panel | Change from baseline after 6 weeks.
  Fasting capillary blood sample for triglycerides and cholesterol
Body mass | Change from baseline after 6 weeks.
  Body mass measured on a scale
Fat mass | Change from baseline after 6 weeks.
  Total and segmental body fat mass measured by DXA
Lean mass | Change from baseline after 6 weeks.
  Total and segmental lean mass measured by DXA
Dietary intake | Change from baseline after 6 weeks.
  Food logs recorded over two week days and one weekend day
Physical activity | Change from baseline after 6 weeks.
  Free-living physical activity assessed over 7 days via combined heart-rate and accelerometry
Depression symptoms | Change from baseline after 6 weeks.
  Symptoms of depression assessed with Beck's Depression Inventory (BDI). The BDI is a 21-item questionnaire that measures total depressive symptoms. Individual item scores range from 0-3. Individual items are then summed to provide a total score, ranging from 0 to 63.

CONTACTS AND LOCATIONS:
Locations (1):
- California State University San Marcos, San Marcos, California, United States

IPD SHARING:
Plan to Share IPD: No